CLINICAL TRIAL: NCT04839003
Title: A Registry to Investigate Real-world Natural History, Impact of Therapies and Patterns of Progression of AL Amyloidosis (ReAL)
Brief Title: A Registry of AL Amyloidosis (ReAL)
Acronym: ReAL
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giovanni Palladini, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: AC-018-IT
Record Dates: First submitted 2021-03-22; First posted 2021-04-09 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-07

CONDITIONS: AL Amyloidosis
Keywords: amyloidosis; prognosis; registry
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — It will be generated a biobank of body fluids (serum, plasma, urine) and relevant cellular (bone marrow and peripheral blood mononuclear cells) and tissue samples (bone marrow, periumbilical fat, possibly other biopsied organs) from patients with AL amyloidosis. We will obtain research samples from diagnostic leftovers of consenting patients at diagnosis and at each subsequent visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this protocol is to generate a large registry of patients with AL amyloidosis.

DETAILED DESCRIPTION:
Thanks to this registry, it will be possible to collect data at diagnosis and during follow up, in order to be able to describe the natural history of AL amyloidosis in a real-world setting and to define and validate prognostic models, response and relapse criteria applicable at any point of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of systemic AL amyloidosis;
2. treatment-naïve (pre-treatment data collected at participating center available for retrospective part);
3. age ≥18 years;
4. ability to understand and willingness to sign an informed consent (patients who already sign informed consent for clinical data to be used in retrospective analyses will be accepted);
5. planned (or ongoing) follow-up at participating center.

Exclusion Criteria:

1. non-AL amyloidosis;
2. previous treatment for AL amyloidosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be entered the database pending on expressing an informed consent of the use of their data for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Creation of a registry of patients with AL amyloidosis | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy